CLINICAL TRIAL: NCT03310541
Title: A Pilot Study of AZD5363 for Patients With Advanced Solid Tumors Harboring Mutations in AKT1, AKT2, or AKT3
Brief Title: AZD5363 in Patients With Advanced Solid Tumors Harboring AKT Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-322
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Prostate Cancer; Advanced Solid Tumors
Keywords: AZD5363; AKT Mutations; 17-322
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — capivasertib; enzalutamide; Fulvestrant

STUDY DESIGN:
Intervention Model Description: This will be an open label, single institution, non-randomized, pilot study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Prostate, Previously treated with Enzalutamide (Experimental): 28-DAY CYCLE AZD5363 400mg PO twice daily for 4 days on, 3 days off, every week + Enzalutamide 160 mg PO once daily
  Interventions: Drug: AZD5363; Drug: Enzalutamide
- ER+ Breast, Previously treated with Fulvestrant (Experimental): 28-DAY CYCLE AZD5363 400mg PO twice daily for 4 days on, 3 days off, every week + Fulvestrant 500mg IM days 1, 15, 29 (cycle 2 day 1) and then every 4 weeks
  Interventions: Drug: AZD5363; Drug: Fulvestrant
- Advanced Solid Tumors (Experimental): 28-DAY CYCLE AZD5363 480mg PO twice daily for 4 days on, 3 days off, every week
  Interventions: Drug: AZD5363

INTERVENTIONS:
Drug: AZD5363 — AZD5363 400mg PO twice daily for 4 days on, 3 days off, every week
Drug: Enzalutamide — Enzalutamide 160 mg PO once daily
  Arms: Prostate, Previously treated with Enzalutamide
Drug: Fulvestrant — 500mg IM days 1, 15, 29 (cycle 2 day 1) and then every 4 weeks
  Arms: ER+ Breast, Previously treated with Fulvestrant

SUMMARY:
This study will test the recommended dose of AZD5363 (recommended from a previous phase 1 study of the drug) in patients with specific AKT mutations. In patients who have ER positive breast cancer with an AKT mutation, they will also be receiving a standard breast cancer drug called fulvestrant that is given as an injection. In patients who have prostate cancer with an AKT mutation, they will also be receiving a standard prostate cancer drug called enzalutamide that is taken orally.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed recurrent or metastatic advanced solid tumor, for which there is no curative-intent treatment option and confirmation of the presence of AKT1, AKT2, or AKT3 mutations detected by the MSK-IMPACT assay platform or other CLIA-approved test
* ER+ breast cancer patients must have received and progressed on Fulvestrant and be post-menopausal
* Prostate cancer patients must have received and progressed on enzalutamide
* Age ≥ 18 years
* ECOG performance status ≤ 2 with no deterioration over the previous 2 weeks
* Life expectancy of ≥ 12 weeks
* Measurable disease as defined by the tumor specific relevant response criteria for the breast and other solid tumor cohorts (measurable disease is not required for enrollment in the prostate cancer cohort):

  * RECIST version 1.1 criteria
  * Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria.
  * RANO criteria
* Females should be using adequate contraceptive measures (see Section 0), should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as:
  * Aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
  * Estradiol, FSH and LH levels in post-menopausal range while receiving LHRH analogues for medical castration in patients with breast cancer.
  * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Male patients should be willing to use barrier contraception (i.e. condoms)

Exclusion Criteria:

* ER+ breast cancer patients harboring the AKT1 E17K mutation (patient population tested in MSK IRB# 14-214, study D3610C00001 part E, ClinicalTrials.gov NCT01226316).
* Diabetes mellitus type 1
* Fasting plasma glucose [fasting is defined as no calorific intake for at least 8 hours]:

  * ≥ 126 mg/dL for those patients without a pre-existing diagnosis of Type 2 diabetes mellitus
  * ≥ 167mg/dL for those patients with a pre-existing diagnosis of Type 2 diabetes mellitus
* Glycosylated haemoglobin (HbA1C) ≥8.0%
* Requirement for insulin for routine diabetic management and control
* Requirement for >2 oral hypoglycaemic medications for routine diabetic management and control
* Treatment with any of the following:

  * Any investigational agents or study drugs from a previous clinical study within 30 days of the first dose of study treatment
  * Any other chemotherapy, immunotherapy or anticancer agents within 3 weeks or 5 half lives, whichever is longer, of the first dose of study treatment, except fulvestrant, enzalutamide or hormonal therapy with LHRH analogues for medical castration in patients with breast or prostate cancer, which are permitted
  * Potent inhibitors or inducers or substrates of CYP3A4 or substrates of CYP2D6 within 2 weeks before the first dose of study treatment (3 weeks for St John"s Wort).
  * Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment
  * Radiotherapy with a wide field of radiation within 4 weeks of the first dose of study treatment
  * Prior ATP-competitive AKT inhibitors
* With the exception of alopecia, any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment
* Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus. Screening for chronic conditions is not required.
* Any of the following cardiac criteria:

  * Resting corrected QT interval (QTc) > 480 msec obtained from electrocardiogram (ECG)
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiogram (ECG) eg, complete left bundle branch block, third degree heart block
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
  * Experience of any of the following procedures or conditions in the preceding 6 months and judged to be clinically significant by Principle Investigator: : coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association (NYHA) Grade ≥2
  * Uncontrolled hypotension - Systolic blood pressure (BP) <90mmHg and/or diastolic BP <50mmHg
  * Left ventricular ejection fraction (LVEF) below lower limit of normal for site.
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

  * Absolute neutrophil count < 1 x 10^9/L
  * Platelet count < 100 x 10^9/L
  * Haemoglobin < 9.0 g/dL
  * ALT > 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases, or >5 times ULN in presence of liver metastases
  * AST > 2.5 times ULN if no demonstrable liver metastases, or >5 times ULN in presence of liver metastases.
  * Total bilirubin > 1.5 times ULN (patients with confirmed Gilbert"s syndrome may be included in the study)
  * Creatinine >1.5 times ULN concurrent with creatinine clearance < 50 ml/min; confirmation of creatinine clearance is only required when creatinine is > 1.5 times ULN
  * Proteinuria 3+ on dipstick analysis or >500 mg/24 hours
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD5363
* History of hypersensitivity to active or inactive excipients of AZD5363, fulvestrant and enzalutamide or drugs with a similar chemical structure or class to these agents.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
number of patients with an objective response rate (ORR) of AZD5363 | 1 year
  A response is defined as any of the following: a response according to RECIST v 1.1, PCWG3 (for patients with measurable visceral and/or nodal disease at baseline) or RANO as applicable or a reduction in the PSA level of 50% or more (for prostate cancer patients without visceral and/or nodal disease at baseline), with a confirmatory assessment at least 4 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Schram, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Shrestha Bhattarai T, Shamu T, Gorelick AN, Chang MT, Chakravarty D, Gavrila EI, Donoghue MTA, Gao J, Patel S, Gao SP, Reynolds MH, Phillips SM, Soumerai T, Abida W, Hyman DM, Schram AM, Solit DB, Smyth LM, Taylor BS. AKT mutant allele-specific activation dictates pharmacologic sensitivities. Nat Commun. 2022 Apr 19;13(1):2111. doi: 10.1038/s41467-022-29638-1. PMID 35440569
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm